CLINICAL TRIAL: NCT06181331
Title: The Effect of a Stepped-care Metacognition-based Intervention on Managing Fear of Cancer Recurrence: Sequential, Multiple Assignment, Randomized Controlled Trial (SMARTs)
Brief Title: The Effect of a Stepped-care Metacognition-based Intervention on Managing Fear of Cancer Recurrence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FCR-SMART
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Fear of Cancer Recurrence
Keywords: Sequential multiple assessment randomized controlled trial; stepped-up care; psychooncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: First stage intervention: We will use a block randomization with randomly permuted block sizes of 2,4, and 6 to ensure close balance of the numbers in each arm. Participants will be randomised to the eConquerFear or eHealthMaintenance
  Second stage intervention for non-respondents: We will use a block randomization with randomly permuted block sizes of 2,4, and 6 to ensure close balance of the numbers in each arm. Participants will be randomised to the augment eConquerFear with eHealthMaintenance (or vice versa) versus switch to supervised, face-to-face ConquerFear intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: he investigator, care provider, investigator and outcomes assessor are masked in terms of not knowing to which condition the participants will be randomized until after the completion of the baseline assessment. The outcomes assessor will break the envelope for the next eligible participant indicating if that participant is to be allocated to intervention or control arms.
  The participants are masked in terms of not knowing that one intervention is hypothesized to yield larger effects than the other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- First stage intervention: eConquerFear (Experimental): Participants in the eConquerFear intervention group will receive six online modules with each containing educational text, illustrative graphics, interactive exercises, and brief videos. Every module will teach a specific topic, such as self-examination and medical surveillance, values-based goal setting, attention training, detached mindfulness, worry management and treatment summary and relapse prevention.
  Interventions: Behavioral: eConquerFear
- First stage intervention: eHealthMaintenance (Active Comparator): Participants in the eHealthMaintenance group will receive six videos, which were designed to provide comprehensive lifestyle guidance (e.g., relaxation techniques, diet and physical activity advices) to help with survivors' maintenance of health in long-term.
  Interventions: Behavioral: eHealthMaintenance
- Second stage intervention: ConquerFear-HK (Experimental): ConquerFear-HK is a culturally adapted, manualized intervention consisting of 6 individual face-to-face sessions over 10 weeks.
  Interventions: Behavioral: ConquerFear
- Second stage intervention: eConquerFear+eHealthMaintenance (Active Comparator): The augmented eConquerFear + eHealthMaintenance intervention is a combined unsupervised, self-guided web-based intervention that consists of 10 weekly online modules covering the content of eConquerFear and eHealthMaintenance interventions.
  Interventions: Behavioral: eConquerFear+eHealthMaintenance

INTERVENTIONS:
Behavioral: eConquerFear — The key goals of this e-intervention are to: (i) teach strategies for controlling worry and excessive threat monitoring; (ii) modify underlying unhelpful MCQ beliefs about worry; (iii) develop appropriate monitoring and screening behaviours, (iv) encourage acceptance of the uncertainty brought about by a cancer diagnosis, and (v) clarify values and encourage engagement in values-based goal setting.
  Arms: First stage intervention: eConquerFear
Behavioral: eHealthMaintenance — eHealthMaintenance is not developed specifically to target fear of cancer recurrence through modifying participants' cognitive beliefs. Participants in this arm will receive 6 videos about relaxation, generic dietary and exercise knowledge.
  Arms: First stage intervention: eHealthMaintenance
Behavioral: ConquerFear — ConquerFear is an intensive version of eConquerFear, which consists of 6 face-to-face therapist-led sessions.
  Arms: Second stage intervention: ConquerFear-HK
Behavioral: eConquerFear+eHealthMaintenance — The combination of eConquerFear and eHealthMaintenance interventions, that consists of 10 weekly online modules.
  Arms: Second stage intervention: eConquerFear+eHealthMaintenance

SUMMARY:
A sequential multiple-assignment randomized controlled trial (SMART) will be used to assess the effect of an adaptive stepped-care intervention on FCR in cancer survivors with subclinical levels of fear of cancer recurrence.

DETAILED DESCRIPTION:
The current SMART trial aims to address the following hypotheses:

Hypothesis 1: It is better to begin adaptive interventions with eConquerFear than with eHealthMaintenance.

Hypothesis 2: Among initial non-respondents, it is better to switch to supervised, face-to-face ConquerFear than to augment eConquerFear with eHealthMaintenance.

Hypothesis 3: eConquerFear + ConquerFear will lead to the greatest reduction in fear of cancer recurrence.

Hypothesis 4: There would be an indirect effect of stepped-care ConquerFear intervention on fear of cancer recurrence through its effect on maladaptive metacognition and cognitive attentional syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese- or Mandarin-speaking Chinese patients diagnosed with curable breast, colorectal, or gynecological cancer, who had completed treatment (except endocrine therapy) within five years, and with a Fear of Cancer Recurrence Inventory-Short Form (FCRI-SF) score of 13 to 21 indicating subclinical FCR will be included.

Exclusion Criteria:

* Patients with metastatic cancer, with a current diagnosis of depression or psychosis, or who are already receiving psychological treatment will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of fear of cancer recurrence (FCR) | baseline (T0), one-month post-intervention (T1), and six-month (T2) post intervention
  The primary outcome is the change in the total score of FCR assessed using the 42-item Fear of Cancer Recurrence Inventory (FCRI). The FCRI measures seven dimensions of FCR: (1) triggers, (2) severity, (3) psychological distress, (4) functional impairment, (5) reassurance, (6) insights, and (7) coping strategies. All items are rated on 5-point Likert scales ranging from 0 (not at all or never) to 4 (a great deal or all the time). Higher scores indicate higher levels of FCR.

SECONDARY OUTCOMES:
Change of metacognitions | baseline (T0), one-month post-intervention (T1), and six-month (T2) post intervention
  Metacognition assessed by the 30-item Metacognitions Questionnaire (MCQ). The MCQ assesses individual differences in metacognitive beliefs, judgements, and monitoring tendencies across five domains: (1) positive beliefs about worry, (2) negative beliefs about thoughts concerning uncontrollability and danger, (3) cognitive confidence, (4) cognitive self-consciousness, and (5) the need to control thoughts. All items are rated on a 4-point Likert scale ranging from 1 (do not agree) to 4 (agree very much). Higher scores indicate higher levels of maladaptive metacognition.
Change of cognitive attentional syndrome | baseline (T0), one-month post-intervention (T1), and six-month (T2) post intervention
  CAS measured by the 16-item Cognitive Attentional Syndrome-1 (CAS-1) questionnaire.The CAS-1 assesses the frequency of engaging in rumination, threat monitoring, and coping behaviors, as well as the level of metacognitive beliefs. Each item is rated on a 9-point Likert scale ranging from 0 to 8, except for items measuring metacognitive beliefs, which are rated on a scale from 0 to 100. Higher scores indicate higher levels of CAS activation.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Lam, PhD, Principal Investigator — School of Public Health, The University of Hong Kong
Locations (1):
- QMh department of surgery, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the PI upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: Information will be available from the PI upon reasonable request. The author to review requests is the PI.